CLINICAL TRIAL: NCT00451152
Title: A Study of the Safety and IOP-Lowering Efficacy of Anecortave Acetate in Patients With Open-Angle Glaucoma
Brief Title: Safety and Efficacy of Anecortave Acetate in Patients With Open-Angle Glaucoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C-06-19
Record Dates: First submitted 2007-03-21; First posted 2007-03-23 (Estimated); Last update posted 2012-11-28 (Estimated); Status verified 2012-05

CONDITIONS: Open-angle Glaucoma
Keywords: glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle; Glaucoma | interventions — anecortave acetate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Anecortave Acetate Depot (Experimental)
  Interventions: Drug: Anecortave Acetate Sterile Suspension, 30 mg/mL
- Anecortave Acetate Vehicle (Placebo Comparator)
  Interventions: Other: Anecortave Acetate Vehicle

INTERVENTIONS:
Drug: Anecortave Acetate Sterile Suspension, 30 mg/mL — Administered by anterior juxtascleral depot (AJD) in study eye, either 0.25 mL or 0.5 mL. One injection, 24 months.
  Arms: Anecortave Acetate Depot
Other: Anecortave Acetate Vehicle — Administered by anterior juxtascleral depot (AJD) in study eye, 0.5 mL. One injection, 24 months.
  Arms: Anecortave Acetate Vehicle

SUMMARY:
The purpose of this study was to evaluate the safety and intraocular pressure (IOP)-lowering efficacy of anecortave acetate for treatment of elevated IOP in patients with open-angle glaucoma.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of open-angle glaucoma;
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Pseudoexfoliation;
* Pigment dispersion component;
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2007-03; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Mean Intraocular Pressure (IOP) | 3 months

SECONDARY OUTCOMES:
Percent Treatment Failures | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Theresa Landry, Ph.D., Study Director — Alcon Research
Locations (1):
- Texas, San Antonio, Texas, United States